CLINICAL TRIAL: NCT07366177
Title: Can the "Face Index"; an Anthropometric Measurement, Predict Difficult Laryngoscopy and Intubation?
Status: Not yet recruiting | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Nilay Tas, Prof. Dr., Ordu University
Other Study IDs: NTasFACE
Record Dates: First submitted 2026-01-18; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Anesthesia Intubation Complication; Laryngoscopy; Intubation; Difficult or Failed; Anesthesia Morbidity
Keywords: Difficult airway, face index, anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Face index — Face index is an anthropometric measurement

SUMMARY:
Patient safety is the cornerstone of anesthetic practice, and maintaining adequate respiration represents its most critical initial step. In situations where spontaneous breathing cannot be sustained-such as during general anesthesia-the airway must be mechanically secured. While simple face masks may be sufficient in some cases, endotracheal intubation remains the most reliable method for airway control in conditions associated with respiratory depression.

Airway management may be challenging due to various patient-related anatomical factors, including facial and mandibular structure, obesity, limited mouth opening, facial hair, sunken cheeks, wide facial morphology, and a short or muscular neck. These challenges are collectively described as difficult ventilation and difficult intubation (cannot ventilate-cannot intubate), which may occur unexpectedly or be anticipated. A difficult airway is defined as difficulty encountered by a trained anesthesiologist in face mask ventilation, tracheal intubation, or both.

Several predictors of difficult airway are widely accepted, such as thyromental and sternomental distances, neck circumference, Mallampati classification, upper lip bite test, mouth opening, and interincisor distance. Thorough preoperative airway evaluation is mandatory, as difficult mask ventilation and failed intubation remain major contributors to anesthesia-related morbidity and mortality. Although numerous studies have examined these predictors, research focusing on facial morphology and anthropometric indices-particularly the face index-is extremely limited.

Facial morphology varies considerably among individuals and can be evaluated anthropometrically using simple, noninvasive tools such as a digital caliper. Anthropometric analysis is commonly applied in forensic medicine and reconstructive surgery but has rarely been incorporated into airway assessment.

This study aims to introduce face index analysis as a novel predictor of difficult airway alongside conventional methods. By evaluating measurements such as trichion-gnathion distance, total facial index, upper facial index, and nasal index, the study investigates whether airway difficulty can be predicted using a single index value. All measurements are standard, noninvasive, and routinely performed during preoperative assessment.

DETAILED DESCRIPTION:
Patient safety is the most critical aspect of anesthetic practice, and the first step in ensuring this safety is the maintenance of adequate respiratory function. Under anesthesia, or in any situation where spontaneous respiration cannot be sustained, the upper and lower airways must be mechanically secured. Airway control can often be achieved using simple face masks; however, in cases of general anesthesia or similar conditions associated with respiratory depression, airway management must be ensured through the more reliable method of endotracheal intubation.

During artificial ventilation, numerous physical characteristics such as facial structure, mandibular anatomy, obesity, limited mouth opening, the presence of a beard, a thin face with sunken cheeks, a wide facial structure, and a short, muscular neck may pose challenges for the anesthesiologist. These situations, defined in the medical literature as "difficult ventilation - difficult intubation" (cannot ventilate - cannot intubate), are not uncommon and may present as either anticipated or unanticipated difficult airways. A difficult airway is defined as a clinical situation in which a trained anesthesiologist experiences difficulty with face mask ventilation, tracheal intubation, or both, due to upper airway conditions (1,2).

Universally accepted predictors of difficult airway among anesthesiologists and the scientific community include physical measurements and classifications such as thyromental distance, sternomental distance, neck circumference, upper lip bite test, Mallampati classification, mandibular length, mouth opening, and interincisor distance (1,3,4). A comprehensive preoperative airway evaluation is both necessary and mandatory during the physical examination of patients scheduled for general anesthesia (5,6). One of the most common-and arguably the most significant-causes of anesthesia-related morbidity and mortality is difficult mask ventilation and failed intubation. In daily anesthetic practice, these classifications are frequently used to reduce the risk of airway difficulty and enhance patient safety, and numerous studies and theses addressing these physical examination criteria are available in the literature.

Despite the abundance of such studies, research evaluating facial morphology and anthropometric measurements-including the "face index"-is almost nonexistent. Facial morphology varies widely among individuals worldwide. It can be analyzed anthropometrically using various measurements and indices, which are currently most commonly applied in fields such as forensic medicine and aesthetic or reconstructive surgery. Anthropometric measurement is a technique that examines metrically definable body characteristics and can be performed easily using a simple measurement tool such as a digital caliper (7).

The primary aim of this study is to introduce a novel perspective on difficult airway assessment by incorporating face index analysis as an additional airway predictor alongside traditional measurement methods that have long been used in anesthesiology. Specifically, the study seeks to determine whether airway difficulty can be predicted using a single index value rather than multiple measurements in patients with different facial morphologies.

Airway management involves sequential steps, beginning with ventilation via a face mask, followed by visualization of the vocal cords (laryngeal inlet and vocal folds) using laryngoscopy, and finally placement of an endotracheal tube into the trachea. Facial measurements may identify physical factors that contribute to difficulty at any of these stages. This study primarily investigates the predictive value of conventional difficult airway assessments in comparison with components of the face index, including trichion-gnathion length (Tri-Gn), total facial index, upper facial index, and nasal index, in determining airway management difficulty.

All measurements employed in this study are standard, noninvasive, and harmless physical examination methods routinely used by anesthesiologists worldwide and are mandatory components of preoperative assessment.

ELIGIBILITY:
Inclusion Criteria:

All adult patients over the age of 18 who have given written consent to undergo elective and/or emergency surgery under general anesthesia and be intubated in the operating rooms of our hospital's main building and annex building

Exclusion Criteria:

Patients with a prior history of difficult airway/difficult intubation, those who have undergone facial, neck, or airway surgery, those with deformities or scars in the facial and neck area due to burns or injuries, those with previous or recent tracheostomy, those with facial deformities due to any cause (congenital or acquired pathologies), and those with communication problems and who are uncooperative during measurements will be excluded from the study. Children and pregnant patients will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over 18 years of age who will undergo general anesthesia and intubation
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Face index and face mask ventilation | 365 days
  Face index is useful measurement about difficult laryngoscopy management in anesthesia

SECONDARY OUTCOMES:
Face index and intubation | 365 days
  Face index is useful measurement about difficult laryngoscopy management in anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Taş, Prof. Dr., Principal Investigator — Ordu University School of Medicine, Türkiye

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Apfelbaum JL, Hagberg CA, Connis RT, Abdelmalak BB, Agarkar M, Dutton RP, Fiadjoe JE, Greif R, Klock PA, Mercier D, Myatra SN, O'Sullivan EP, Rosenblatt WH, Sorbello M, Tung A. 2022 American Society of Anesthesiologists Practice Guidelines for Management of the Difficult Airway. Anesthesiology. 2022 Jan 1;136(1):31-81. doi: 10.1097/ALN.0000000000004002. PMID 34762729
- [Result] Coskun A, Duzgun SA, Bozer M, Akinci OF, Uzunkoy A. Modified technique for correction of gynaecomastia. Eur J Surg. 2001 Nov;167(11):822-4. doi: 10.1080/11024150152717643. PMID 11848235
- [Result] Jackson JS, Rondeau B. Mallampati Score. 2025 Jul 7. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK585119/ PMID 36256766
- [Result] Chow HH, Tolle KM, Roe DJ, Elsberry V, Chen H. Application of neural networks to population pharmacokinetic data analysis. J Pharm Sci. 1997 Jul;86(7):840-5. doi: 10.1021/js9604016. PMID 9232526
- [Result] Garber DA, Beverley SM, Coen DM. Demonstration of circularization of herpes simplex virus DNA following infection using pulsed field gel electrophoresis. Virology. 1993 Nov;197(1):459-62. doi: 10.1006/viro.1993.1612. PMID 8212585
- [Result] Vidon N, Palma R, Bernier JJ. [Water-electrolyte movements along the human intestine in diarrhea induced by mannitol]. Gastroenterol Clin Biol. 1983 Jan;7(1):23-9. No abstract available. French. PMID 6404686